CLINICAL TRIAL: NCT02484105
Title: Comforting Conversation During Colonoscopy: A Randomised Controlled Trial on Patient Satisfaction
Brief Title: Comforting Conversation During Colonoscopy: A Trial on Patient Satisfaction
Acronym: ComConEndo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeppe Thue Jensen (Other)
Responsible Party: Sponsor-Investigator, Jeppe Thue Jensen, MD, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-15001924
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comforting Conversation (Experimental): Conversation according to the initital qualitative study.
  Interventions: Behavioral: Comforting Conversation; Behavioral: Standard Communication
- Standard Communication (Active Comparator): Standard information prior to and during endoscopy.
  Interventions: Behavioral: Standard Communication

INTERVENTIONS:
Behavioral: Comforting Conversation — Pain management, distraction, diversion, empathy. Dependent on qualitative study results.
  Arms: Comforting Conversation
Behavioral: Standard Communication — Information on procedure type, duration, findings, key landmarks, possibility of analgesic treatment, pause in procedure.

SUMMARY:
Does comforting conversation during colonoscopy improve on patient satisfaction, compliance and pain management.

DETAILED DESCRIPTION:
Does comforting conversation during colonoscopy improve on patient satisfaction, compliance and pain management. A randomized controlled trial on comforting conversation or standard communication during colonoscopy. Using a mixed methods model, a qualitative study will be conducted to clarify what patients deem as important or effective conversation during colonoscopy. A randomized controlled trial will hereafter be conducted, where the results from the initial study will be utilized in the conversation during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Colonoscopy
* Written informed content

Exclusion Criteria:

* ASA Class 4 or higher
* BMI 40 or higher
* Analgesics taken prior to procedure
* Pregnancy or breast feeding
* Allergy to Fentanyl/Midazolam
* Daily consumption of opioids
* Unable to complete questionnaire

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | on average 20 minutes after completed colonoscopy.
  Questionnaire with 5 point Likert like scale

SECONDARY OUTCOMES:
Per-procedural Pain management | From inclusion to completed procedure. On average 45 minutes from first to last measurement.
  Pain/discomfort prior to-, every 5. minutes and post-procedure with patients using the Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy, Gastrounit, Herlev Hospital, Herlev, Region H, Denmark